CLINICAL TRIAL: NCT00340678
Title: Renoprotection in Early Diabetic Nephropathy in Pima Indians
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 999995037; OH95-DK-N037 (Other: NIH/NIDDK)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2013-10

CONDITIONS: Diabetic Nephropathy
Keywords: Angiotensin II Receptor Antagonist; Therapeutic Trial; Glomerular Filtration Rate; Kidney Biopsy; Non-Insulin Dependent Diabetes Mellitus
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normoalbuminuria Losartan (Experimental): Subjects with normal urinary albumin excretion were treated with losartan began at 50 mg daily, with the dose increasing to 100 mg daily after 1 week if symptomatic hypotension did not develop.
  Interventions: Drug: Losartan
- Normoalbuminuria Placebo (Placebo Comparator): Subjects with normal urinary albumin excretion were treated with placebo corresponding to each dose of losartan.
  Interventions: Drug: Placebo
- Microalbuminuria Losartan (Experimental): Subjects with microalbuminuria were treated with losartan began at 50 mg daily, with the dose increasing to 100 mg daily after 1 week if symptomatic hypotension did not develop.
  Interventions: Drug: Losartan
- Microalbuminuria Placebo (Placebo Comparator): Subjects with Microalbuminuria were treated with placebo corresponding to each dose of losartan.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Treatment with losartan began at 50 mg daily, with the dose increasing to 100 mg daily after 1 week if symptomatic hypotension did not develop.
  Other Names: Cozaar; MK-954; DuP 753
  Arms: Microalbuminuria Losartan; Normoalbuminuria Losartan
Drug: Placebo — Treatment with placebo corresponding to each dose of losartan.
  Arms: Microalbuminuria Placebo; Normoalbuminuria Placebo

SUMMARY:
This investigation is a randomized, double-blinded, placebo-controlled clinical trial in adult diabetic Pima Indians with normal urinary albumin excretion (albumin-to-creatinine ration less than 30 mg/g) or microalbuminuria (albumin-to-creatinine ration = 30-299 mg/g) to test the hypothesis that blockade of the renin-angiotensin system with the angiotensin receptor blocker (ARB) losartan can prevent or further attenuate the development and progression of early diabetic nephropathy in subjects with type 2 diabetes mellitus who are receiving standard diabetes care.

One hundred seventy subjects were recruited for the study, all of whom had type 2 diabetes for at least 5 years, serum creatinine concentrations less than 1.4 mg/dl, and no evidence of non-diabetic renal diseases. Ninety-two of the subjects had normal urinary albumin excretion at baseline and other 78 had microalbuminuria. Subjects in each albumin excretion group were randomized to treatment with either the angiotensin II receptor antagonist, losartan, or placebo. Measurements of glomerular filtration rate (GFR), renal plasma flow (RPF) and fractional clearances of albumin and IgG will be made initially, at one month, and at 12-month intervals from baseline thereafter. A kidney biopsy was performed after six years in 111 subjects. Morphometric analysis of renal biopsies was used to determine differences in glomerular structure between treatment groups.

DETAILED DESCRIPTION:
This investigation is a randomized, double-blinded, placebo-controlled clinical trial in adult diabetic Pima Indians with normal urinary albumin excretion (albumin-to-creatinine ratio < 30 mg/g) or microalbuminuria (albumin-to-creatinine ratio = 30-299 mg/g) to test the hypothesis that blockade of the renin-angiotensin system with the angiotensin receptor blocker (ARB) losartan can prevent or further attenuate the development and progression of early diabetic nephropathy in subjects with type 2 diabetes mellitus who are receiving standard diabetes care.

One hundred seventy subjects were recruited for the study, all of whom had type 2 diabetes for at least 5 years, serum creatinine concentrations < 1.4 mg/dl, and no evidence of non-diabetic renal diseases. Ninety-two of the subjects had normal urinary albumin excretion at baseline and the other 78 had microalbuminuria. Subjects in each albumin excretion group were randomized to treatment with either the angiotensin II receptor antagonist, losartan, or placebo. Measurements of glomerular filtration rate (GFR), renal plasma flow (RPF) and fractional clearances of albumin and immunoglobulin G (IgG) were made initially, at one month, and at 12-month intervals from baseline thereafter. A kidney biopsy was be performed after six years in 111 subjects. Morphometric analysis of renal biopsies was used to determine differences in glomerular structure between treatment groups.

The major outcome measure was a decline in GFR to less than or equal to 60 ml/min or to half the baseline value in subjects that enter the study with a GFR of < 120 ml/min. Other measures of renoprotection were assessed, including group differences in 1) change in albumin excretion, 2) change in serum creatinine concentration, and 3) glomerular morphology in all subjects as outlined above.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers from the Gila River Indian Community who meet the eligibility criteria will be invited to participate.

To be eligible for participation in the study, subjects must meet the following criteria:

* Aged 18-65.
* Diagnosis of type 2 diabetes greater than or equal to 5 years.
* Serum creatinine concentration less than to 1.4 mg/dl.
* Serum potassium concentration less than or equal to 5.5 milliequivalents (mEq)/L.
* At least 2 of 3 weekly screening urinary albumin-to-creatinine ratios less than 300 mg/g. All screening tests are to be within 3 months of enrollment.
* Willingness, after receiving a thorough explanation of the study, to participate.

EXCLUSION CRITERIA:

Subjects will be excluded for the following reasons:

* Clinically significant disorders of the liver, cardiovascular disease, cerebrovascular disease, peripheral vascular disease, pulmonary diseases, renal-urinary disorders, gastrointestinal disorders, or hematocrit levels less than or equal to 30 percent in women or less than or equal to 35 percent in men.
* Renovascular or malignant hypertension; uncontrolled hypertension despite treatment with three antihypertensive drugs; or hypertension that is being treated with antihypertensive medicines and the primary care physician or the patient refuses to adopt the blood pressure treatment regimen outlined in the study protocol.
* Hematuria of unknown etiology.
* Chronic debilitating disorders with or without treatment that would interfere with the assessment of kidney function or that might reduce the chances of survival for a sufficient length of time to evaluate efficacy of treatment.
* Currently receiving a drug regimen that includes: steroids, immunosuppressants, or investigational new drugs.
* Pregnancy. Women of childbearing potential must have a negative pregnancy test prior to entry and every three months during the study.
* Evidence of inability to empty the bladder.
* Hypersensitivity to angiotensin-converting enzyme inhibitors (ACEi), ARBs, or iodine.
* Bleeding disorders, since kidney biopsies could not be performed safely in these individuals.
* Massive obesity with body mass index greater than or equal to 45 kg/m(2).
* Non-diabetic renal disease.
* Conditions that are likely to interfere with informed consent or compliance with the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 1995-08; Primary Completion 2012-05 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Nelson, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Zatz R, Meyer TW, Rennke HG, Brenner BM. Predominance of hemodynamic rather than metabolic factors in the pathogenesis of diabetic glomerulopathy. Proc Natl Acad Sci U S A. 1985 Sep;82(17):5963-7. doi: 10.1073/pnas.82.17.5963. PMID 3862110
- [Background] Zatz R, Dunn BR, Meyer TW, Anderson S, Rennke HG, Brenner BM. Prevention of diabetic glomerulopathy by pharmacological amelioration of glomerular capillary hypertension. J Clin Invest. 1986 Jun;77(6):1925-30. doi: 10.1172/JCI112521. PMID 3011862
- [Background] Anderson S, Rennke HG, Garcia DL, Brenner BM. Short and long term effects of antihypertensive therapy in the diabetic rat. Kidney Int. 1989 Oct;36(4):526-36. doi: 10.1038/ki.1989.227. PMID 2681929
- [Result] Weil EJ, Fufaa G, Jones LI, Lovato T, Lemley KV, Hanson RL, Knowler WC, Bennett PH, Yee B, Myers BD, Nelson RG. Effect of losartan on prevention and progression of early diabetic nephropathy in American Indians with type 2 diabetes. Diabetes. 2013 Sep;62(9):3224-31. doi: 10.2337/db12-1512. Epub 2013 Apr 1. PMID 23545707
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Fort PE, Rajendiran TM, Soni T, Byun J, Shan Y, Looker HC, Nelson RG, Kretzler M, Michailidis G, Roger JE, Gardner TW, Abcouwer SF, Pennathur S, Afshinnia F. Diminished retinal complex lipid synthesis and impaired fatty acid beta-oxidation associated with human diabetic retinopathy. JCI Insight. 2021 Oct 8;6(19):e152109. doi: 10.1172/jci.insight.152109. PMID 34437304
- [Derived] Reynolds EL, Akinci G, Banerjee M, Looker HC, Patterson A, Nelson RG, Feldman EL, Callaghan BC. The determinants of complication trajectories in American Indians with type 2 diabetes. JCI Insight. 2021 May 24;6(10):e146849. doi: 10.1172/jci.insight.146849. PMID 34027894
- [Derived] Afshinnia F, Nair V, Lin J, Rajendiran TM, Soni T, Byun J, Sharma K, Fort PE, Gardner TW, Looker HC, Nelson RG, Brosius FC, Feldman EL, Michailidis G, Kretzler M, Pennathur S. Increased lipogenesis and impaired beta-oxidation predict type 2 diabetic kidney disease progression in American Indians. JCI Insight. 2019 Nov 1;4(21):e130317. doi: 10.1172/jci.insight.130317. PMID 31573977
- [Derived] Tanamas SK, Saulnier PJ, Fufaa GD, Wheelock KM, Weil EJ, Hanson RL, Knowler WC, Bennett PH, Nelson RG. Long-term Effect of Losartan on Kidney Disease in American Indians With Type 2 Diabetes: A Follow-up Analysis of a Randomized Clinical Trial. Diabetes Care. 2016 Nov;39(11):2004-2010. doi: 10.2337/dc16-0795. Epub 2016 Sep 9. PMID 27612501
- [Derived] Weil EJ, Lemley KV, Mason CC, Yee B, Jones LI, Blouch K, Lovato T, Richardson M, Myers BD, Nelson RG. Podocyte detachment and reduced glomerular capillary endothelial fenestration promote kidney disease in type 2 diabetic nephropathy. Kidney Int. 2012 Nov;82(9):1010-7. doi: 10.1038/ki.2012.234. Epub 2012 Jun 20. PMID 22718189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between 1996 and 2001, the last biopsy was performed in 2007, and morphometric evaluation was completed in 2012.
Pre-assignment Details: Of 313 patients with type 2 diabetes who were screened, 79 were ineligible, 50 declined to participate, and 14 had other reasons that prevented participation despite meeting eligibility requirements.
Period: Overall Study
Arm/Group | Normoalbuminuria Losartan | Normoalbuminuria Placebo | Microalbuminuria Losartan | Microalbuminuria Placebo
Started | 46 | 46 | 39 | 39
Completed | 45 | 46 | 39 | 39
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Of 170 subjects enrolled, one lost follow up. So all analysis was performed based on 169 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normoalbuminuria Losartan | Normoalbuminuria Placebo | Microalbuminuria Losartan | Microalbuminuria Placebo | Total
Number analyzed (Participants) | 46 | 46 | 39 | 39 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (10.6) | 41.9 (11.7) | 41.8 (8.9) | 42.3 (10.9) | 41.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 28 | 27 | 124
  Male | 10 | 13 | 11 | 12 | 46
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 39 | 39 | 170
Diabetes duration [Mean (Standard Deviation); unit: years] | 8.8 (4.7) | 10.4 (6.0) | 10.3 (5.2) | 14.1 (8.4) | 10.8 (6.2)
BMI [Mean (Standard Deviation); unit: kg/(m^2)] — Body Mass Index obtained by measuring the participant's height in meters and weight in kilograms.
  kg/(m^2) | 37.4 (8.8) | 36.6 (8.0) | 34.6 (9.1) | 33.8 (7.2) | 35.7 (8.3)
Blood pressure, systolic [Mean (Standard Deviation); unit: mmHg] | 115 (11) | 118 (14) | 118 (15) | 123 (13) | 118 (13)
Blood pressure, diastolic [Mean (Standard Deviation); unit: mmHg] | 75 (7) | 75 (7) | 77 (9) | 77 (7) | 76 (7)
Blood pressure, mean [Mean (Standard Deviation); unit: mmHg] | 88 (7) | 89 (9) | 90 (10) | 92 (8) | 90 (9)
HbA1c [Mean (Standard Deviation); unit: %] — Glycosylated hemoglobin is an integrated measure of glycemic control that reflects an average glycemic level over the past 3 months.
  % | 9.2 (2.0) | 8.1 (2.2) | 9.5 (2.3) | 10.3 (2.1) | 9.2 (2.1)
Glomerular filtration rate (GFR) [Mean (Standard Deviation); unit: mL/min] — Glomerular filtration rate was measured by the urinary clearance of iothalamate.
  mL/min | 171 (38) | 152 (40) | 166 (43) | 168 (43) | 164 (41)
Urinary albumin to creatinine ratio [Median (Inter-Quartile Range); unit: mg/g] | 15 [10 to 23] | 14 [9 to 26] | 66 [39 to 205] | 80 [46 to 165] | 47 [9 to 205]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Decline in GFR
Description: Participants were monitored for up to 6 years. This is the number of participants who had a decline in GFR to less than or equal to 60 ml/min or to half the baseline value in subjects that enter the study with a GFR of less than 120 ml/min during the time of observation.
Time Frame: Up to 6 years
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Normoalbuminuria Losartan | Normoalbuminuria Placebo | Microalbuminuria Losartan | Microalbuminuria Placebo
Number analyzed (Participants) | 45 | 46 | 39 | 39
participants | 2 | 2 | 1 | 4

2. Secondary Outcome: Glomerular Volume
Time Frame: 6 years after first treatment
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: *10^6 cubic microns
Arm/Group | Normoalbuminuria Losartan | Normoalbuminuria Placebo | Microalbuminuria Losartan | Microalbuminuria Placebo
Number analyzed (Participants) | 45 | 46 | 39 | 39
*10^6 cubic microns | 5.4 (1.8) | 5.6 (1.1) | 6.4 (2.3) | 7.0 (3.0)

ADVERSE EVENTS:
Groups:
- Losartan: Subjects received losartan
- Placebo: Subjects received placebo
Arm/Group | Losartan | Placebo
Serious Adverse Events (participants affected / at risk) | 3/84 | 6/85
Other Adverse Events (participants affected / at risk) | 1/84 | 0/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=84) | Placebo (N=85)
Death from coronary artery disease (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Death from leukemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Death from hepatocellular carcinoma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Death from alcoholic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Death from automobile accident (Social circumstances) | 0 (0) | 2 (2)
Death from multiple myeloma (General disorders) | 1 (1) | 0 (0)
Death from bleeding gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=84) | Placebo (N=85)
Urethral obstruction after kidney biopsy (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes